CLINICAL TRIAL: NCT05683990
Title: DiaPrecise, A Phase II Open Label Study to Evaluate the Safety and Feasibility of Intralymphatic Administration of Diamyd® in Individuals at Risk for Type 1 Diabetes Carrying the HLA DR3-DQ2 Haplotype
Brief Title: Study to Evaluate the Safety and Feasibility of Diamyd® in Individuals at Risk for Type 1 Diabetes
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Diamyd Medical AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DiaPrecise (D/P2/22/8)
Record Dates: First submitted 2022-12-20; First posted 2023-01-13 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus, Type 1; Autoimmune Diseases; Prevention
Keywords: HLA DR3-DQ2; Metabolic Disease; Autoimmune Diabetes; Vitamin D; Immune System Diseases; GAD65; Residual c-peptide; T1D; Type 1 Diabetes; Diamyd; retogatein
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Autoimmune Diseases; Metabolic Diseases; Immune System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): 2 injections of Diamyd
  Interventions: Drug: Diamyd
- Arm 2 (Experimental): 3 injections of Diamyd
  Interventions: Drug: Diamyd

INTERVENTIONS:
Drug: Diamyd — 4 μg (0.1 mL) of Diamyd administered 1 month apart.

SUMMARY:
A 2-arm randomized Phase II Open Label Study to evaluate the safety and feasibility of intralymphatic administration of Diamyd® (Diamyd) also known as retogatein in individuals at risk of Type 1 diabetes carrying the HLA DR3-DQ2 haplotype.

DETAILED DESCRIPTION:
The trial is a 2-arm, randomized, open label clinical trial in individuals aged 8 - <18 years with HLA DR3-DQ2 and multiple islet autoantibodies (Stage 1 or Stage 2) at increased risk for T1D. At baseline eligible individuals at risk of T1D will be randomized 1:1 into 2 or 3 injections of Diamyd® also known as retogatein administered into an inguinal lymph node. Subjects will be followed for a total of 12 months post-enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent/assent from the individual and the individual's parents or caretaker(s) according to local regulations.
2. Males and females aged ≥8 and <18 years old at the time of Screening.
3. Possess the HLA DR3-DQ2 haplotype.
4. Seropositive for GADA and at least one additional T1D-associated autoantibody (IA-2A, ZnT8A or IAA).

Exclusion Criteria:

1. Diagnosis of T1D (stage 3 T1D, according to the American Diabetes Association [ADA] classification).
2. Fasting glucose > 7 mmol/L (126 mg/dl), 2-hour-OGTT plasma glucose > 11.1 mmol/L (200 mg/dL) or HbA1c > 6.5% (48 mmol/mol) at the screening Visit.
3. Treatment with any anti-diabetic medication, including the use of external insulin.
4. Participation in any other clinical trial testing pharmaceutical treatments.
5. Recent (past 12 months) or current treatment with immunosuppressant therapy, including chronic use of glucocorticoid therapy. Inhaled, topical, and intranasal steroid use is acceptable. Short courses (e.g., ≤5 days) of oral or intra-articular injections of steroids will be permitted on trial.
6. History of hyperparathyroidism, hypercalcemia and/or nephrolithiasis, unless appropriately treated, or any other contraindication to use of Vitamin D.
7. History of epilepsy, serious head trauma or cerebrovascular accident, or clinical features of continuous motor unit activity in proximal muscles
8. Any clinically significant history of an acute reaction to a vaccine or its constituents (e.g., Alhydrogel) or lidocaine (local anesthetic)
9. Any acute or chronic skin infection or condition that would preclude intralymphatic injection.
10. Treatment with any (live or inactive) vaccine, including influenza vaccine and Coronavirus Disease 2019 (COVID-19) vaccine, within 4 weeks prior to planned first dose of study drug; or planned treatment with any vaccine up to 4 weeks after the last injection with study drug.
11. Ongoing diagnosed post-COVID19 syndrome.
12. Known diagnosis of human immunodeficiency virus (HIV), hepatitis B or hepatitis C infection. Individuals with previous hepatitis C infection that is now cured may be eligible.
13. Any clinically significant concomitant medical condition, including but not limited to other autoimmune diseases, cardiovascular, gastrointestinal, hematological, immune, renal including a history of renal transplantation or neurological that in the opinion of the investigator would interfere with trial participation or procedures. Celiac disease with adequate diet as well as stable autoimmune thyroiditis will be permitted.
14. Any clinically significant abnormal findings detected during Screening that might jeopardize the individual's safety or ability to complete the trial.
15. Females who are lactating or pregnant (for females who have started menstruating the possibility of pregnancy must be excluded by urine βHCG onsite prior to the study drug administration).
16. Males or females not willing to use adequate contraception, if sexually active, until 90 days after the last Diamyd administration. Adequate contraception is as follows:

For females of childbearing potential (FOCBP)

1. oral (except low-dose gestagen (lynestrenol and norestisteron)), injectable, or implanted hormonal contraceptives
2. intrauterine device
3. intrauterine system (for example, progestin-releasing coil)
4. refraining from heterosexual intercourse if that is the preferred and usual lifestyle of the subject.

For sexually active males

1. condom
2. Abstinence from heterosexual intercourse if that is the preferred and usual lifestyle of the subject.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-07-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of AEs (including Injection site reactions) and SAEs | From screening to 12 months.
Number of Clinically Significant Abnormal Results from Physical examinations, including neurological and Vital Signs assessments | From screening to 12 months.
Number of Clinically Significant Abnormal Results From Laboratory measurements, including hematology, clinical chemistry, metabolic status parameters (fasting C-peptide, HbA1c, fasting glucose) and urine analysis | From screening to 12 months.

SECONDARY OUTCOMES:
Stage progression | From screening to 12 months.
  Number of individuals progressing from stage 1 to stage 2 and from stage 2 to stage 3.
T1D diagnosis | From screening to 12 months.
  Time to T1D diagnosis.
Time to stage progression | From screening to 12 months.
  Time from stage 1 to stage 2 and time from stage 2 to stage 3.
OGTT stimulated C-peptide | From screening to 12 months.
  Change in C-peptide /insulin /glucose (Area Under the Curve [AUC]mean 0-120 min) during a 2-hour Oral Glucose Tolerance Test (OGTT) from screening to 12 months.
Change in Hemoglobin A1c (HbA1c) | From baseline to 12 months.
  Change in Hemoglobin A1c (HbA1c) from baseline to 12 months.
Change in time in glycemic target range | From screening to 12 months.
  Change in time in glycemic target range 3.9 to 10 mmol/L (70 to 180 mg/dL) and 3.9 to 7.8 mmol/L (70 to 140 mg/dL) evaluated from continuous glucose monitoring (CGM) data from screening to 12 months.
Change in time in range > 13.9 mmol/L | From screening to 12 months.
  Change in time in range > 13.9 mmol/L (> 250 mg/dL) evaluated from CGM data from screening to 12 months.
Change in time in range > 10 mmol/L | From screening to 12 months.
  Change in time in range > 10 mmol/L (> 180 mg/dL) evaluated from CGM data from screening to 12 months.
Change in time in range > 7.8 mmol/L | From screening to 12 months.
  Change in time in range > 7.8 mmol/L (> 140 mg/dL) evaluated from CGM data from screening to 12 months.
Change in glycemic variation | From screening to 12 months.
  Change in glycemic variation (Coefficient of variation [CV], SD) evaluated from CGM data from screening to 12 months.
Variables that indicate effects on the immune system | From baseline to 12 months.
  Variables that indicate effects on the immune system such as the concentration of serum autoantibodies.

CONTACTS AND LOCATIONS:
Locations (1):
- Lund University/CRC, Skåne University Hospital,, Malmo, Sweden